CLINICAL TRIAL: NCT04577183
Title: A Prospective, Open Label, Multicenter Trial for Evaluating the Efficacy of Treating and Managing Wounds in Elderly Population in Specialized Nursing Facilities Using RedDress Wound Care System (RD1)
Brief Title: A Prospective, Open Label, Multicenter Trial for Evaluating the Efficacy of Treating and Managing Wounds in Elderly Population in Specialized Nursing Facilities Using RD1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: operational challenges
Sponsor: RedDress Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD004
Record Dates: First submitted 2019-03-20; First posted 2020-10-06 (Actual); Results first posted 2021-05-13 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Foot Ulcer; Pressure Ulcer; Venous Leg Ulcer; Trauma Injury; Skin Tear; Chronic Ulcer
MeSH Terms: conditions — Diabetic Foot; Pressure Ulcer; Varicose Ulcer; Accidental Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- RD1 System (Experimental): The RD1 is created by drawing the patient's blood with the use of citrate anticoagulant. The anticoagulant allows the clot to form later in a controlled fashion-citrate is a widely used anticoagulant. The blood is then placed in the clotting tray (within few minutes) and the coagulation is facilitated by adding calcium and kaolin (insoluble aluminum silicate). The forming clot assumes the shape of the tray containing it, and can then be applied to the wound, and then covered with primary and secondary dressings.
  Interventions: Device: RD1 System

INTERVENTIONS:
Device: RD1 System — The RD1 is created by drawing the patient's blood with the use of citrate anticoagulant. The anticoagulant allows the clot to form later in a controlled fashion-citrate is a widely used anticoagulant. The blood is then placed in the clotting tray (within few minutes) and the coagulation is facilitated by adding calcium and kaolin (insoluble aluminum silicate). The forming clot assumes the shape of the tray containing it, and can then be applied to the wound, and then covered with primary and secondary dressings.

SUMMARY:
The study is a prospective, single arm, multicenter efficacy study, consisting of 60 subjects who will complete the study (note: if any patients are lost to follow-up or withdrawn, enrollment will increase to compensate for loss of these subjects). The subjects will receive up to 16 RD1 applications. In case of complete healing, subject will be called for one confirmatory visit two weeks later or before discharge from the SNF (the earlier of the two). Subject data will be kept in each site's records.

All diabetic subjects' glycemic management will be performed by a qualified physician. All subjects will have wound care specialist or wound surgeon or dermatologist involved in their wound care

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years of age
* Patient with a wound deemed suitable for treatment with RD1
* Ulcer free of clinical signs of infection.
* Post-debridement, ulcer free of necrotic tissue.
* For foot ulcers, Subject has adequate vascular perfusion of the affected limb, as defined by - Ankle-Brachial Index (ABI) ≥ 0.65 and ≤ 1.2
* HbA1c ≤ 12.0% (diabetic patients)
* Subject or legal authorized representative must be willing to comply with the protocol including having blood drawn to create the RD1.
* Female subjects who are capable of conceiving must use an acceptable form of contraception in order to participate in the study (acceptable forms of contraception include condoms for males and contraceptive pills or IUDs for women).

Exclusion Criteria:

* If ulcer area decreases by ≥ 30% during the initial 2-week screening (± 2 days) and standard of care phase, or if the ulcer area increases ≥ 30%,
* Presence of active underlying osteomyelitis.
* Patient with a proven sepsis established by a blood culture in the past 2 weeks, or confirmed active infection likely to interfere with trial, such as urine tract infection
* Known malignancy in the reference wound bed or margins of the wound
* Exposure of blood vessels or organs at the base of the reference wound
* History of alcohol or substance abuse, within the previous 2 months
* Subject has participated in another clinical trial involving a device or a systemically administered investigational study drug or treatment within 30 days of day 0 visit.
* Subject is currently receiving (i.e., within the past 30 days) or scheduled to receive a medication or treatment which, in the opinion of the Investigator, is known to interfere with, or affect the rate and quality of, wound healing (e.g., systemic steroids (more than 10mg per day), immunosuppressive therapy, autoimmune disease therapy, cytostatic therapy within the past 12 months, dialysis, radiation therapy to the ulcer area, vascular surgery, angioplasty or thrombolysis).
* Subject has been treated with wound dressings that include growth factors, engineered tissues or skin substitutes within 30 days of randomization or is scheduled to receive during the study.
* Subject has been treated with hyperbaric oxygen within 5 days of screening or is scheduled to receive during the study.
* Wound on a patient who has a life expectancy of less than 6 months.
* Cannot withdraw blood in the required amount technically.
* Known coagulation problems, abnormal thrombocytes level or if heparin is given intravenously. Patients who are taking orally Coumadin, Aspirin, or Plavix (clopidogrel) will not be excluded.
* Hemoglobin anemia (< 9 g/dL).
* Subject has an infectious disease, such as Acquired Immune Deficiency Disease (AIDS) or HIV, Hepatitis C, Hepatitis B, Human T-lymphotropic virus or Syphilis
* Women who are pregnant or currently breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnyview Nursing & Rehabilitation Center, Butler, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RD1 System
Started | 13
Completed | 7
Not Completed | 6
Not completed — Death | 1
Not completed — Withdrawal by Subject | 3
Not completed — Early termination | 2

BASELINE CHARACTERISTICS:
Arm/Group | RD1 System
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reduction in Wound Size
Description: Numer of patients showed Percent of wound reduction from baseline to end of treatment in the intent to treat (ITT) population
Time Frame: 16 weeks
Population: Number of patients showed Percent of wound reduction in the intent to treat (ITT) population
Measure: Number; unit: participants with Wound Size reduction
Arm/Group | RD1 System
Number analyzed (Participants) | 13
participants with Wound Size reduction | 7

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | RD1 System
All-Cause Mortality (participants affected / at risk) | 1/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RD1 System (N=13)
Death (Cardiac disorders) | 1 (1) — Heart failure
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RD1 System (N=13)
Multiple fluid filled blisters to left lower extrimity (Musculoskeletal and connective tissue disorders) | 1 (1)
Open area on right upper shin (Musculoskeletal and connective tissue disorders) | 1 (1)
Cellulitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Skin tear (Skin and subcutaneous tissue disorders) | 1 (5)
New ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Infection to study ulcer (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
The study had a Statistical Analysis Plan in progress that wasn't finalized. Due to the small group size, conclusions could be made without conducting statistics for the study population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT04577183/Prot_001.pdf